CLINICAL TRIAL: NCT03856827
Title: A Phase 1 Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of IW-6463 When Administered to Healthy Volunteers as Single Ascending Doses, as Multiple Ascending Doses, and Under Fed Versus Fasting Conditions
Brief Title: A Study of IW-6463 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tisento Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: C6463-101; CY6463 (Other: Cyclerion Therapeutics)
Record Dates: First submitted 2019-02-20; First posted 2019-02-27 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Other

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IW-6463 (Experimental): IW-6463 tablets administered orally as single ascending doses, multiple ascending daily doses, and single doses with or without food
  Interventions: Drug: IW-6463
- Placebo (Placebo Comparator): Matching placebo tablets administered orally
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: IW-6463 — IW-6463 Tablet
  Other Names: CY6463; zagociguat
  Arms: IW-6463
Drug: Matching Placebo — Matching Placebo Tablet
  Arms: Placebo

SUMMARY:
Stage 1: To assess the safety and tolerability of single-ascending-dose levels of IW-6463 tablets when administered orally to healthy subjects

Stage 2: To assess the safety and tolerability of multiple-ascending-dose levels of IW-6463 tablets administered orally to healthy subjects

Stage 3: To assess the safety and tolerability of a single dose of IW-6463 when administered to health subjects in fed vs fasted states and explore the effects of food on IW-6463 pharmacokinetics (PK)

ELIGIBILITY:
Inclusion Criteria:

* Subject is an ambulatory adult between 18 and 64 years old at the screening visit with the exception of the elderly cohort, who must be 65 years or older at the screening visit.
* Subject is in good health and has no clinically significant findings on physical examination
* Women of reproductive potential must have a negative pregnancy test at the time of check-in and must agree to use protocol-specified contraception throughout the duration of the study and for 3 months after the final dose of study drug
* Men must agree to use protocol-specified contraception and also to not donate sperm throughout the study and for 3 months after the final dose of study drug
* Other inclusion criteria per protocol

Exclusion Criteria:

* Any active or unstable clinically significant medical condition
* Use of any prescribed or non-prescribed medication
* Other exclusion criteria per protocol

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
After single ascending doses, number of subjects with treatment-emergent adverse events (TEAEs) in the IW-6463 dose-level cohorts vs the (pooled) placebo group. | Up to 9 days
After multiple ascending doses, number of subjects with TEAEs in the IW-6463 dose-level cohorts vs the (pooled) placebo group. | Up to 32 days
After a single dose, number of subjects with TEAEs in the fed vs fasted dosing period | Up to 28 days
Plasma concentration of IW-6463 after single-dose administration under fed vs fasted conditions | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Chad Glasser, PharmD, Study Director — Cyclerion Therapeutics, Inc; Geert J Groeneveld, MSc, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands